CLINICAL TRIAL: NCT03110302
Title: In-Home Exposure Therapy for Veterans With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-12- 1-0614
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Telehealth; Video teleconferencing; In home therapy; Prolonged Exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Office-based telehealth (OBT) (Active Comparator): Veterans come to a VA clinic and meet with a therapist via telehealth, using videoconferencing technology
  Interventions: Behavioral: Prolonged exposure
- Home-based telehealth (HBT) (Active Comparator): Veterans stay at home and meet with the therapist via telehealth, using videoconferencing technology
  Interventions: Behavioral: Prolonged exposure
- In home, in person (IHIP) (Experimental): Therapist goes to the Veterans' homes to provide the psychotherapy
  Interventions: Behavioral: Prolonged exposure

INTERVENTIONS:
Behavioral: Prolonged exposure — PE is a manualized treatment developed by Dr. Edna Foa and her colleagues. In all three treatment modalities, 7-15 weekly, 90 minute individual sessions of PE will be provided. PE is based on emotional processing theory, which proposes that avoidance and negative thoughts about the self and the world maintain PTSD symptoms over time. According to emotional processing theory, effective treatment requires repeated activation of the trauma memory (as through memory and in vivo exposure) and incorporation of corrective information into the trauma fear structure. PE has several primary components: (1) psychoeducation about PTSD and avoidance; (2) imaginal exposure with processing, wherein the participant describes the traumatic memory aloud many times and discusses it with the therapist afterward; and (3) in-vivo exposure, wherein the participant engages in feared, but safe, activities that have been avoided since the traumatic event (e.g., crowded places, driving).
  Other Names: PE

SUMMARY:
This study examines clinical and process outcomes following variable length prolonged exposure (PE) for posttraumatic stress disorder (PTSD) delivered by one of three treatment modalities: home-based telehealth (HBT), office-based telehealth (OBT), or in-home-in-person (IHIP).

DETAILED DESCRIPTION:
This study will provide a certain type of exposure therapy, called prolonged exposure therapy (PE), to military Veterans with Post Traumatic Stress Disorder (PTSD). One hundred and seventy-five Veterans will participate in the study. The main study goal is to compare PE conducted in three different ways: (1) PE that is office-based (OB; Veterans come to a VA clinic and meet with a therapist via telehealth, using videoconferencing technology), (2) PE delivered via home-based telehealth (HBT; Veterans stay at home and meet with the therapist via telehealth, using videoconferencing technology), and (3) PE delivered in home, in person (IHIP; the therapist goes to the Veterans' homes to provide the psychotherapy). Symptoms of PTSD, depression, and anxiety will be examined at pre-treatment, post-treatment and at six-month follow up to determine if symptoms change over time. Study hypotheses state that the IHIP approach, compared to the other two approaches, will be more effective at reducing the PTSD symptoms experienced by these Veterans because it will help Veterans attend each session and complete the therapy "homework" assigned by the therapists (such as doing feared, but safe, activities around the house or the neighborhood). However, the delivery of IHIP may cost more than the delivery of PE via the other modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Military Veterans enrolled in a program at VASDHS;
2. primary diagnosis of PTSD as a consequence of any index traumatic event. The diagnosis will include a clear memory of the traumatic event and the 17 other core symptoms of PTSD from the DSM-IV. Note that comorbid mood and anxiety disorders are expected and will be permitted (to maximize generalizability) if PTSD symptoms are judged to be predominant based on primacy and severity of symptoms. The proposed treatment often concurrently ameliorates depression and anxiety symptoms;
3. age 18 or older; and
4. Primary residence within 35 miles of the center point of La Jolla, CA center (to make therapist travel to home sites feasible for this project). This will include the major cities of San Diego, Chula Vista (23 miles Southeast; 30 minutes), La Mesa (19 miles East; 25 minutes), Coronado (18 miles South; 30 minutes), Oceanside (36 miles Southeast; 39 minutes), Escondido (27 miles northeast; 35 minutes) and San Ysidro (28 miles South; 32 minutes).

Exclusion Criteria:

1. unmanaged dementia, psychosis or manic episodes in past year (assessed by phone screen, chart review, and clinician judgment);
2. substance or alcohol dependence in past 60 days (as assessed by the Alcohol Use Disorders Identification Test [AUDIT]);
3. concurrent psychotherapies targeting PTSD (Veterans who are engaged in treatment for non PTSD symptoms, such as 12-step programs for substance problems or couples therapy for relationship issues, will remain eligible); and
4. severe physical disease or disorder (e.g., cardiovascular or respiratory disease; severe impairments in speech, vision, or hearing) that would make it difficult to ensure regular attendance at psychotherapy sessions or would significantly impede learning (as assessed during phone screen discussion with potential participants). Potential participants who have had changes in the type and dosage of psychotropic medications in the preceding 60 days will be asked to wait until their medication regimen has stabilized to minimize treatment confounds. Psychotropic medication use will also be monitored to determine whether random assignment to treatment conditions resulted in unequal rates of use. As recommended by Bradley and colleagues, individuals with suicidal ideation will not be excluded from the study a priori, but rather suicidal urges or plans will be assessed throughout the study and appropriately addressed (by intervention or referral). The depression measure (the BDI-II) assesses suicidality explicitly (item 9). Dr. Thorp has extensive experience working with suicidal individuals and teaching crisis management skills, and the other study therapists will be trained in these skills as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | From baseline to 9 months
  The CAPS is a clinician-administered interview that assesses PTSD severity and diagnostic threshold. CAPS questions are designed to assess DSM-5 PTSD diagnostic criteria. CAPS has become the "gold standard" semistructured interview for assessing PTSD in the general population.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory (BDI-II) | From baseline to 9 months
  The BDI is a well-established, 21-item self-report inventory designed to measure depressive symptomatology, including suicidality.
Change in PTSD Checklist (PCL-5) | From baseline to 9 months
  The PCL-5 is a gold-standard self-report questionnaire designed to assess PTSD symptom severity; there are 20 questions.
Change in Client Satisfaction Questionnaire (CSQ) - Short form | From baseline to 3 months
  This well-validated questionnaire consists of 8 items rated on a 5-point Likert scale ranging from "Not at all" to "Very much" and one free response question. The CSQ is designed to measure patient satisfaction with interpersonal and communication behaviors.
Change in Therapist Satisfaction Questionnaire (TSQ) | From baseline to 3 months
  The TSQ is a validated instrument filled out by the therapist and used to measure provider satisfaction with therapy. This questionnaire consists of 20 items that are rated on a 5-point likert scale raning from "Strongly agree" to "Strongly disagree."
Change in Working Alliance Inventory - Short form (WAI-S) | From baseline to 3 months
  The WAI measures therapeutic alliance between the therapist and patient. Both the patient and the therapist fill out the WAI. This 12-item inventory has 3 subscales: (1) Goals (agreement about therapy goals), (2) Tasks (agreement about issues to be worked on), and (3) Bonds (comfort level between participant and therapist).

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Morland, PsyD, Principal Investigator — VA San Diego and University of California, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morland LA, Mackintosh MA, Glassman LH, Wells SY, Thorp SR, Rauch SAM, Cunningham PB, Tuerk PW, Grubbs KM, Golshan S, Sohn MJ, Acierno R. Home-based delivery of variable length prolonged exposure therapy: A comparison of clinical efficacy between service modalities. Depress Anxiety. 2020 Apr;37(4):346-355. doi: 10.1002/da.22979. Epub 2019 Dec 24. PMID 31872563